CLINICAL TRIAL: NCT06238726
Title: Nudging Patients to Increase Shingles Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Massachusetts Institute of Technology (Other); National Bureau of Economic Research, Inc. (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor & Director of Decision Sciences, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-1504
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Shingles; Vaccination Behavior; Behavior, Health
MeSH Terms: conditions — Herpes Zoster; Health Behavior

STUDY DESIGN:
Masking Description: Although patients will not be explicitly informed of which arm they were randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Passive control (No Intervention): Patients in this arm will not be sent any messages.
- Active control (Active Comparator): Patients in this arm will be sent messages encouraging them to ask about Shingrix at their upcoming appointment.
  Interventions: Behavioral: Reminder
- High risk (Experimental): Patients in this arm will be sent messages informing them that they are at high risk for shingles because they are ages 50+, and encouraging them to ask about Shingrix at their upcoming appointment.
  Interventions: Behavioral: Reminder
- Multi-fact (Experimental): Patients in this arm will be sent messages with facts about shingles and Shingrix, and encouraging them to ask about Shingrix at their upcoming appointment.
  Interventions: Behavioral: Reminder
- High risk + multi-fact (Experimental): Patients in this arm will be sent messages informing them that they are at high risk for shingles because they are ages 50+, with additional facts about shingles and Shingrix, and encouraging them to ask about Shingrix at their upcoming appointment.
  Interventions: Behavioral: Reminder

INTERVENTIONS:
Behavioral: Reminder — Shingrix messages via SMS, patient portal, email, and/or another modality
  Arms: Active control; High risk; High risk + multi-fact; Multi-fact

SUMMARY:
The purpose of this study is to test whether messages encouraging patients to ask about a Shingrix vaccine at an upcoming appointment will increase Shingrix vaccination rates. The study will also test which of several message versions is most effective.

DETAILED DESCRIPTION:
Shingles is a painful disease caused by reactivation of the varicella zoster (chickenpox) virus. About a third of adults in the US will develop shingles in their lifetime, with the highest prevalence in adults ages 50 and older. Roughly one in ten patients with shingles develops complications that can lead to long-term pain and inflammation). Shingrix, a two-shot vaccine series, is highly effective at preventing shingles and is recommended by the CDC for all adults ages 50 and over.

The present study will test whether sending patients messages encouraging them to ask about Shingrix at an upcoming primary care appointment increases vaccination rate relative to Passive Control (no messages). Additionally, four message arms will vary as a function of risk (message includes or does not include a statement telling patient they are at high risk for shingles because they are age 50+) and facts (message includes or does not include several facts about shingles and Shingrix), with the no-high-risk, no-facts arm designated as the Active Control arm.

Message arms will be crossed with two additional randomized variables: number of messages (2 messages or 3 messages) and cost information (the presence or absence of information about the cost of Shingrix in the final message).

Enrollment timing will vary by insurance group. Enrollment will begin with patients who have a Geisinger Health Plan (GHP) membership that allows them to get Shingrix at no cost (this includes the vast majority of GHP members), because existing data allow the study team to easily identify these patients and inform them about their Shingrix coverage in cost messages. Enrollment for patients who are not GHP members (and the few patients with a GHP plan that is not Shingrix eligible) will begin following the development of an automated internal process that will allow cost messages to include information about patients' individualized Shingrix insurance benefits. Alternatively, if development is delayed approximately 2 months or longer from the launch of enrollment for GHP members, the study team may decide in collaboration with Geisinger leadership to begin enrolling patients without GHP using a generic cost message (e.g., "Most patients can get Shingrix at no cost").

Enrollment for each insurance group (GHP members, non-GHP members) will begin with a 2-week pilot period, with a limited number of new patients (e.g., 100 to 200) enrolled per day in that insurance group (these patients will be randomly selected from the eligible patients). During the pilot period, the study team will communicate frequently with clinical partners to ensure there are no issues before full rollout. If issues arise, the pilot period may be extended. If the pilot period does not result in any changes to outreach, or involves only trivial changes, patients enrolled in the pilot period will be included in analysis. If there are more substantive changes to the outreach following the pilot period, patients enrolled during that period will be excluded from analysis.

Once full rollout occurs, enrollment for each insurance group will last for 1 year. Study enrollment will be complete 1 year following full rollout for non-GHP members.

Anticipated enrollment is at least 50,000.

UPDATE ON 4/15/24: Following a recent review of clinical operational workflows, clinical stakeholders determined that the copays estimated through the automated process will typically not be applicable to non-GHP members. Therefore, in the coming weeks, text messaging to eligible non-GHP members will begin, with a generic cost message for those randomized to be sent a cost message.

UPDATE ON 8/6/24: From September through December 2024, a flu vaccination text message nudge campaign will be running at Geisinger for similar appointments as this shingles vaccination study. Clinical leadership has decided that patients should only receive nudge messages about one vaccine per appointment, and that flu shot messages should be prioritized during flu season. Instead of pausing shingles vaccination messages entirely during the flu campaign, the team will enroll patients in the shingles study if they have already gotten a flu vaccine this flu season according to the EHR. The inclusion criteria are now updated to reflect this change.

The original plan (described above) was to run for one year for each insurance group, as described above, with at least 50,000 patients enrolled during this time. Because there is less certainty that enrollment will reach (or surpass) 50,000 patients during the predefined time frame, the study will end for GHP patients after enrollment reaches 50,000 patients. For non-GHP patients, the study will run for 5 additional weeks before stopping completely, because non-GHP launch occurred 5 weeks after GHP launch. This way, the study length will be the same for both insurance groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 50+
* Has not received any doses of the Shingrix vaccine according to the Geisinger EHR
* Has a non-acute in-person Geisinger primary care appointment in a department that stocks Shingrix scheduled with enough time to be randomized

Exclusion Criteria:

* Cannot be contacted via the communication modality being used in the study (e.g., patient portal, SMS), e.g., due to insufficient/missing contact information in the EHR or because they opted out
* Patient does not have an approved insurance on file for Shingrix outreach for their appointment type or department
* Appointment type or department not approved for outreach by Geisinger leadership at the time of outreach
* While a separate flu vaccination nudge campaign is running (approximately from September through December, 2024), patients will be excluded if they have not received a flu shot in the 2024-25 flu season according to the EHR. Such patients will be eligible for inclusion again as soon as the flu vaccination campaign ends.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50786 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
First Shingrix vaccination | 3 days after enrollment
  Received a first Shingrix vaccination on the appointment date (y/n)

OTHER OUTCOMES:
First Shingrix vaccination | In the 10 days following enrollment
  Received a first Shingrix vaccination in the 10 days following enrollment (y/n)
Attended scheduled appointment | 3 days after enrollment
  Attended the target Shingrix-eligible appointment (y/n)
First Shingrix vaccination | In the 14 months following enrollment
  Received a first Shingrix vaccination in the 14 months following enrollment (y/n)
Time to first Shingrix vaccination | In the 14 months following enrollment
  Number of days between enrollment and first Shingrix vaccination
Completion of Shingrix series | In the 14 months following enrollment
  Completed Shingrix vaccination series by getting a second Shingrix vaccination (y/n)
Time to completion of Shingrix series | In the 14 months following enrollment
  Number of days between first and second Shingrix vaccination
Shingles diagnosis | In the 14 months following enrollment
  Diagnosed with shingles (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

REFERENCES:
- See also: CDC (2022). About Shingles (Herpes Zoster). — https://www.cdc.gov/shingles/about/index.html

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT06238726/SAP_001.pdf